Official title:comparative study of nonintubated uniport thoracoscopic surgery using thoracic paravertebral nerve block versus intercostal nerve block for peripheral solitary pulmonary

nodule patients

NCT number:03086213

Document date:April 7,2020

Informed consent form

Updated:April 7,2020

Purpose of the study

The purpose of this study is to compare with the safety and efficient on paravertebral nerve block for the nonintubated uniport thoracoscopic surgery for patients with peripheral solitary pulmonarynodules

Who sponsor this study?

This study is sponsored by the thoracic surgical department of Shenzhenthird people'shospital. Adverse effects during the study There is conventional procedure of regional anesthesia such as paravertebral nerve block guided by ultrasound or intercostal nerve block by thoracoscopy ,so it is determined the total protocols of this study is safe for the eligible subjects. However, there is somewhat uncomfortable for the medical serve during the operation.

The amount of drawing blood for every subject is approximately 10ml.

Can you delete the study at any time?

Ok, if you want to exit the study due to any reason, you can do that .

What is benefical for the eligiable subjects?

There is 100 RMB of additional fee for the subjects of the study. he information of the subjects for admitting the study is confidentiality, so you can not afraid about the reveal yourself privacy.

Who can you communicate with?

If you have any question, you can communicate with the principal of this study, whose moble is 13823135410

Patient signature

date

Doctor

signature at